CLINICAL TRIAL: NCT00600002
Title: A Phase I Clinical Trial of GM-CSF Administration as a Biological Adjuvant in Clinically-Staged, Resectable Pancreatic Adenocarcinoma
Brief Title: Administration as a Biological Adjuvant in Clinically-Staged, Resectable Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Edward Nelson (Other)
Responsible Party: Sponsor-Investigator, Edward Nelson, Dr. Edward Nelson, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 02-69; 2003-2972 (Other: University of California, Irvine)
Record Dates: First submitted 2008-01-17; First posted 2008-01-24 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Resectable Pancreatic Adenocarcinoma; Pancreatic Cancer
Keywords: GM-CSF; Leukine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-CSF (Experimental): Cohort 1: 50 ug/m2 given Intravenous. Cohort 2: 150 ug/m2 given Intravenous. Cohort 3: 250 ug/m2 given Intravenous. Cohort 4: 0 ug/m2 and vehicle (normal saline) given Intra-tumoral. Cohort 5: 50 ug/m2 given Intra-tumoral. Cohort 6: 150 ug/m2 given Intra-tumoral. Cohort 7: 250 ug/m2 given Intra-tumoral.
  Interventions: Biological: GM-CSF

INTERVENTIONS:
Biological: GM-CSF — Cohort 1: 50 ug/m2 given Intravenous. Cohort 2: 150 ug/m2 given Intravenous. Cohort 3: 250 ug/m2 given Intravenous. Cohort 4: 0 ug/m2 and vehicle (normal saline) given Intra-tumoral. Cohort 5: 50 ug/m2 given Intra-tumoral. Cohort 6: 150 ug/m2 given Intra-tumoral. Cohort 7: 250 ug/m2 given Intra-tumoral.

SUMMARY:
The application of immunotherapeutic strategies that target the most potent antigen presenting cell, the dendritic cell (DC), are likely to substantially increase the magnitude of the anti-tumor immune response. Although there are issues of activation state and antigen load, mechanisms to increase the number of DCs available to the immune system are among the first steps in development of affective DC based immunotherapeutic strategies. The Central Hypothesis of our study is: Administration of Granulocyte Macrophage Colony Stimulating Factor (GM-CSF) to patients with pancreatic adenocarcinoma will result in enhance recruitment of DCs to the sentinel lymph node, into the peripheral blood, and/or tumor site. We propose performing a phase I, dose escalation, clinical trial of systemic and intra-tumoral GM-CSF administration for the treatment of pancreatic adenocarcinoma. This trial will be designed to assess toxicity and immunologic effects, principally dendritic cell recruitment. Patients with resectable pancreatic adenocarcinoma by clinical staging criteria will be eligible for enrollment.

The trial we propose is a phase I clinical trial of the addition of GM-CSF as a biological adjuvant to standard care for patients with potentially resectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological proven adenocarcinoma of the pancreas with potentially resectable disease based upon clinical staging.
* Expected survival must be greater than three (3) months.
* A Karnofsky Performance Status (KPS) must be 70 or greater.
* Patients must be >18 years of age. Because Leukine® is a "Pregnancy Category C" drug, female patients must be not be lactating and must be surgically sterile (via hysterectomy or bilateral tubal ligation), postmenopausal, or using acceptable methods of contraception if they are of child bearing potential. Female patients of childbearing potential must also have a negative serum pregnancy test.
* Patients must be able to understand and sign an informed consent form, which must comply with U.S. regulations (U.S. 21 Code of Federal Regulations (CFR) 50) and International Conference on Harmonisation (ICH) guidelines. Availability of alternative curative treatment must be fully explained to the patient and documented in the informed consent form.
* Eligible patients must meet the following laboratory parameters:
* White blood cell (WBC) >3,000/mm3
* Platelets >100,000/mm3
* Hct >33% or Hgb >10.5 gm/dL
* Prothrombin time (PT) within 3 seconds of control
* Serum creatinine <1.5 mg/dL
* Serum calcium <11.0 mg/dL
* Serum Amylase < 2 times the upper limit of normal
* Negative HIV-Ag and HIV-Ab

Exclusion Criteria:

* Patients who have undergone previous treatment with a biological response modifier (interferons, interleukins) or prior immunotherapy within four (4) weeks of study enrollment.
* Patients currently requiring corticosteroids, under immune suppression for any reason including an organ allograft.
* Patients with known contraindications to analgesia or endoscopy.
* Patients with unstable cardiovascular disease (Class IV cardiovascular disease according to the New York Heart Association's functional criteria).
* Patients with any acute or chronic illness as judged clinically significant by the Investigators.
* Patients who have received prior chemotherapy or radiation therapy to the thorax within four (4) weeks of enrollment.
* Prior surgery within 30 days of execution of the informed consent form.
* Persistent fever greater than 39 degrees Celsius unless clinical assessment attributes the etiology to be tumor.
* Primary malignancy (present or remote) of sites other than the pancreas, except for the basal cell epithelioma of the skin.
* Use of investigational drugs within 30 days of execution of the informed consent form.
* Clinically significant (symptomatic) third space fluid collection (i.e.: ascites, pleural effusion).
* Patients with a diagnosis of an autoimmune state, or any psychiatric illness that in the opinion of the Investigators would compromise treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Evaluate toxicity, dendritic cell recruitment, and immune parameters | 2 years

SECONDARY OUTCOMES:
Evaluate patient survival | 2 years
Evaluate progression free survival | 2 years
Evaluate time to treatment failure | 2 years
Evaluate quality of life | 2 years
Evaluate biochemical markers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward L Nelson, M.D., Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States